CLINICAL TRIAL: NCT01726595
Title: Ultrasound Measurement of Reactive Hyperemia in Critical Care: Prognostic and Pathophysiologic Significance
Brief Title: Ultrasound Measurement of Reactive Hyperemia in Critical Care
Acronym: URHC
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Anthony P. Pietropaoli, Professor of Medicine, University of Rochester
Other Study IDs: 00030546
Record Dates: First submitted 2012-07-06; First posted 2012-11-15 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Severe Sepsis; Critical Illness
Keywords: critical care; severe sepsis; microvascular function; ultrasound
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine specimens will be obtained within 48 hours of diagnosis of severe sepsis or severe non-infectious systemic inflammatory response syndrome. Subsequent blood and urine samples will be obtained 3-5 days after the first set of samples, within 48 hours of ICU discharge, and within 48 hours of hospital discharge. Samples will analyzed immediately or stored at -80 degrees celsius until use.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- severe sepsis: Patients with severe sepsis or septic shock
- non-infected critically ill: Patients with severe non-infectious systemic inflammatory response syndrome
- healthy: healthy volunteers

SUMMARY:
The investigators hypothesize that doctors and nurses can undergo a brief period of training and then use ultrasound to accurately measure blood flow in a forearm artery after a brief period when this flow is interrupted with a blood pressure cuff, a measurement the investigators call reactive hyperemia. Reactive hyperemia indicates whether the small blood vessels in the body are healthy -- lower reactive hyperemia indicates worse small blood vessel function. When measured by experienced ultrasound experts, low reactive hyperemia strongly predicts death in critically ill patients with infection (severe sepsis).

The investigators are conducting this study to determine if doctors and nurses, without specific pre-existing expertise in ultrasound, can be trained to make these measurements accurately. If so, the investigators will prove that these measurements can be applied reliably in real-world practice.

The investigators also hypothesize that reactive hyperemia predict the outcomes of illness not just in patients with severe infection, but in other critically ill patients as well.

Finally, the investigators hypothesize that reduced blood flow after blood pressure cuff occlusion is linked with other abnormalities of blood, previously identified in critically ill patients. For example, red blood cells from patients with severe sepsis have been shown to be stiffer than normal, so they are less able to flow along the small blood vessel passages of the body. Red blood cells become stiffer when there is a certain type of stress in the body known as "oxidative stress."

If the investigators show that low reactive hyperemia, stiff red blood cells, and oxidative stress are linked, the investigators hope to develop new treatments that reduce oxidative stress, reduce the stiffness of red blood cells, and in turn improve reactive hyperemia. Improvements in reactive hyperemia indicate improvements in small blood vessel function. Better small blood vessel function means better delivery of oxygen throughout the body. The investigators believe that this will improve outcomes for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to University of Rochester Medical Center ICU services with 2 of the 4 systemic inflammatory response syndrome (SIRS) criteria and acute organ dysfunction will be considered for enrollment.
* Healthy control subjects >= 18 years of age will be recruited from the University and Rochester region at large.

Exclusion Criteria

* Critically ill patients:

  1. Refusal of patient or designated surrogate decision-maker to provide written informed consent, or inability to obtain consent within 48 hours of diagnosis
  2. Attending physician refusal
  3. Hematocrit (Hct) < 21%
  4. Acute bleeding requiring PRBC transfusion
  5. History of chronic, dialysis dependent renal failure
  6. End-stage liver disease and Child-Pugh Grade C
  7. History of organ, bone marrow, or stem cell transplant
  8. Pregnancy
  9. Cardiac surgery (including ventricular assist device prior to first sample collection)
  10. Do not resuscitate at screening or plans for withdrawal of life support imminent
  11. Suicide attempt or intentional drug overdose;
  12. Jehovah's witness
* Healthy Control subjects:

  1. Absent doppler signal in brachial or radial arteries.
  2. Asymmetric cyanosis, poor capillary refill or cold temperature
  3. Known venous thrombosis or there is asymmetric swelling (arm circumference > 2 inches larger than opposite side).
  4. Evidence of inflammation or impaired skin integrity of the involved limb.
  5. History of surgery involving the blood or lymphatic vessels of this limb, including axillary lymph node dissection, will preclude this testing.
  6. History of Anemia or G6PD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill Patients:
  Patients admitted to University of Rochester Medical Center ICU services with 2 of the 4 systemic inflammatory response syndrome (SIRS) criteria and acute organ dysfunction will be considered for enrollment.
  Healthy Control subjects:
  Healthy control subjects >= 18 years of age will be recruited from the University and Rochester region at large.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
hospital mortality | vital status at hospital discharge, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P. Pietropaoli, M.D., M.P.H., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Wexler O, Morgan MA, Gough MS, Steinmetz SD, Mack CM, Darling DC, Doolin KP, Apostolakos MJ, Graves BT, Frampton MW, Chen X, Pietropaoli AP. Brachial artery reactivity in patients with severe sepsis: an observational study. Crit Care. 2012 Dec 12;16(2):R38. doi: 10.1186/cc11223. PMID 22390813